CLINICAL TRIAL: NCT05724979
Title: The Natural Sperm Selection in Intracytoplasmic Sperm Injection (ICSI)
Brief Title: Outcome of Using Sperm Bound to the Zona Pellucida of Immature Oocytes for Intracytoplasmic Sperm Injection (ICSI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hager Ali Muhammed Abu Elmagd, Embryologist, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP-bound sperm technique
Record Dates: First submitted 2022-12-11; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Intracytoplasmic Sperm Injection; Infertility, Male
Keywords: Intracytoplasmic sperm injection (ICSI); zona pellucida (ZP); natural sperm selection; Sperm-oocyte interaction; ZP-bound sperm
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Oocytes of the control group were injected with conventionally selected spermatozoa based on sperm morphology and motility after being processed density gradient centrifugation
- treatment (Experimental): ZP-bound sperm were selected from the surface of the immature oocytes through the use of a microneedle (Sunlight Medical, Jacksonville, FL, USA) and transferred in a 10 % polyvinylpyrrolidone (PVP) solution (SAGE, USA), immobilized, and then used to inject sibling MII oocytes
  Interventions: Other: ZP-binding

INTERVENTIONS:
Other: ZP-binding — The ZP is selective with regard to binding and can bind to normally functioning sperm, especially those with a normal acrosomal region
  Arms: treatment

SUMMARY:
In vivo, the zona pellucida (ZP) of the oocyte can bind to normally functional sperm. The ZP-sperm interaction is one of the final steps of natural selection during their journey in the female reproductive tract. In the current study, we evaluated the ability of the ZP of immature oocytes to harvest the fittest sperm. We compared the embryological outcomes of intracytoplasmic sperm injection (ICSI) using conventionally selected sperm (control group) and ZP-bound sperm (intervention group). Our results showed no statistically significant superiority for the ZP binding technique over the conventional sperm selection with respect to the rates of fertilization and cleavage. However; the rates of blastocyst formation and high-quality blastocysts were significantly improved in the intervention group compare to the control group. These findings imply that the proposed technique can serve as a cost-effective and natural sperm selection method that has the potential to enhance the embryological and clinical outcomes of intracytoplasmic sperm injection (ICSI).

DETAILED DESCRIPTION:
The quality of the selected sperm used for intracytoplasmic sperm injection (ICSI) plays a detrimental role in embryonic quality and development. In in vitro fertilization (IVF) and during the sperm journey through the female reproductive tract in vivo, sperm interact with the zona pellucida (ZP) of the oocyte, which is the last stage of sperm selection before entering the oocyte. The ZP is selective with regard to binding and can bind to normally functioning sperm, especially those with a normal acrosomal region. According to Liu et al., only 14 % of the motile spermatozoa in fertile men can bind to the ZP. Only those spermatozoa with relatively normal size and shape of the acrosomal region and those with no or low Deoxyribonucleic acid (DNA) fragmentation can bind to and the ZP and fuse with the plasma membrane of the oocyte (oolemma) and thus are capable of fertilizing the oocyte. Human sperm vary in size, morphology, DNA integrity, motility, membrane composition, etc., and this can be observed even in the same ejaculate. It is a given fact that thorough sperm selection procedures befall spermatozoa in the female genital tract to filter superior sperm and allow only a small subpopulation of spermatozoa with superior quality to reach the site of fertilization where another sperm selection occurs (i.e. ZP interaction).

The sperm traits that make in vitro fertilization effective are still debated. ICSI is now the standard practice for most Assisted Reproduction technologies (ART) centers worldwide and accounts for approximately 70% of all in vitro fertilization. The routine selection of spermatozoa for ICSI depends on an embryologist subjectively selecting sperm based on their motility and morphology. It is done after an analysis of the seminal fluid, which is a poor predictive tool of male fertility and does not express the fertilization capacity of the sperm. It had assumed that mimicking the natural sperm selection may improve the quality of selected spermatozoa and hence, the clinical outcomes of ICSI. Ideally, a sperm selection method that reduces the number of spermatozoa to a subpopulation with potentially the highest quality can improve fertilization and embryo quality and development and subsequent clinical outcomes of ICSI.

Over the years, several sperm selection techniques have been developed for ICSI. However, these techniques were designed to select sperm based on a single sperm parameter (i.e. motility, density, sedimentation, nuclear integrity, etc.) and ignoring other sperm parameters related to the capability to fertilize the oocyte. Sperm selection techniques such as swim-up, microfluidics, and density gradient centrifugation yield a population of highly motile sperm but fail to mimic the rigorous natural sperm selection that considers other sperm parameters. Moreover, most of these methods require centrifugation which may negatively affect the paternal DNA and reduces the quality of sperm by increasing reactive oxygen species. Following these techniques, an embryologist has to subjectively select sperm based on their motility and morphology, which does not guarantee DNA integrity and is potentially time-consuming.

One of the developed sperm selection methods to relatively duplicate the natural selection is the hyaluronic acid (HA) binding-based Physiological intracytoplasmic sperm injection (PICSI)® dishes. The cumulus oophorus layer surrounding the oocyte consists mainly of HA. However, there is conflicting data on the results using PICSI dishes. Moreover, sperm-ZP binding comprises parameters other than HA that are not featured in PICSI dishes.

Sperm-oocyte interaction is a multi-step process involving physical and molecular interactions. It involves a complex and complementary receptor/ligand-based process between the surface proteins expressed on the ZP and the sperm. Research has unveiled several ZP protein candidates postulated to play a role in binding sperm. The main protein of these is the zona pellucida glycoprotein 3 (ZP3), whose O-linked oligosaccharide chains bind to an acrosome-intact sperm and induce an acrosomal reaction.

The study consisted of 20 patients undergoing ICSI

Our inclusion criteria included:

Female age ≤ 38 years old. Male age ≤ 50 years old. Having at least one immature oocyte (i.e. germinal vesicle (GV) or Metaphase I (MI) oocyte) for incubation with sperm to preserve mature ones for ICSI.

At least 10% sperm motility and thus testicular sperm samples were excluded. The patients were selected based on the percentage of DNA fragmentation and only those with ≤ 20% were recruited. Sibling oocytes were randomly divided into a control and an intervention group. Oocytes of the control group were injected with conventionally selected spermatozoa based on sperm morphology and motility. For the intervention group, one immature oocyte was incubated with a calculated volume of the processed semen with a concentration of 500,000 motile sperm/oocyte in a Carbon dioxide (CO2) incubator for 10 to 30 minutes and then checked for bound sperm under an inverted microscope. Only bound sperm with normal morphology were selected and transferred to a Polyvinylpyrrolidone (PVP) drop for immobilization and then injected into the cytoplasm of the MII oocytes of the intervention groups.

Clinical manipulations

1. Controlled ovarian hyperstimulation (COH): All female patients were injected daily with a subcutaneous follicle-stimulating hormone (Gn, Gonal-F, Merck Serono, United States of America) from the 3rd to the 5th day of the menstrual cycle.

The follicles were checked for reaching the appropriate diameter (i.e. 18-20 mm) and for their number using an ultrasound device. If two or more follicles reached the appropriate diameter, a trigger (human chorionic gonadotropin (hCG)), (Ovitrelle®; Merck Serono, Switzerland) was administered intramuscularly to encourage final maturation and induce ovulation.

2-Sperm preparation: After male couples had been instructed to abstain from sexual activities for 1 to 7 days, Semen samples were collected by masturbation. Samples were placed at room temperature on warm plates or incubators at 37ºc until they were liquefied and the time of liquefaction was recorded.

Both macroscopic and microscopic assessments were performed using the 2010 World Health Organization (WHO) manual as a reference. Then, samples were treated by one of the following techniques depending on the male factor:

For the treatment groups, a specific volume of the prepared semen was co-incubated with an immature oocyte in an injection dish containing 10 µl micro drops of global media (LifeGlobal, Europe) with 3 ml of sterile equilibrated mineral oil overlay at 37 °C with 6 % CO2 for 10- 30 minutes. The volume according to the equation:

x=(pellet volume x 0.5 x 100)/(motility x count (after processing)) 3-Oocyte retrieval: Oocyte retrieval was performed approximately 36 hours following the administration of the ovulation trigger. Under ultrasound guidance, a single lumen gauge needle (Reproline, Germany) had been used to aspirate the follicles for fast oocyte pick-up with a negative pressure of 115-120 mm Hg. At the same time, the follicular fluid had been collected in round bottom sterile 14 ml falcon tubes. Under a stereo microscope, the oocyte-cumulus complexes (COCs) were identified, washed, and transferred into fertilizing global total media (LifeGlobal, Europe) and incubated at 6% CO2 at 37°C until denudation.

4- Oocyte denudation and scoring: The COCs were denudated by placing them into a 100 µ1 drop of buffered media containing hyaluronidase enzyme 80 IU/ml (LifeGlobal, Europe) for 30 to 45 seconds. Then the oocytes were gently aspirated in and out by a sterile stripper pipette resulting in the removal of the coronal cells (25). Following that, a global total w/HEPES Buffer (LifeGlobal, Europe) was used to wash the denudated oocytes. An inverted microscope equipped with automatic manipulators, Narishige, hot stage, and Hoffman optics (Olympus 1x71) was used for assessing the oocytes' maturity. The oocyte maturation assessment was as follows: mature oocytes in the metaphase II (MII) characterized by the extrusion of the polar body, and immature oocytes were either in the germinal vesicle phase (GV) characterized by a centrally located germinal vesicle or in the Metaphase I (MI) characterized by the absence of both the polar body and the germinal vesicle. Mature oocytes were then incubated in a culture medium in a Labotect incubator with 6% Co2 at 37 ºC until the time of the intracytoplasmic sperm injection. In contrast, sibling immature oocytes were incubated in a culture medium (50 µ) with a 5000 concentration of spermatozoa/oocyte and placed in the Labotect incubator for 10-30 minutes till the time of sperm selection.

5- ICSI: Mature oocytes were placed in 10 µl micro drops of the global total w/HEPES Buffer (LifeGlobal, Europe) covered with 3ml of pure equilibrated mineral oil for ICSI.

In the control group, each MII oocyte was injected with a conventionally selected sperm based on morphology and motility after being processed by density gradient centrifugation(DGC). However, in the treatment groups, ZP-bound sperm were selected from the surface of the immature oocytes through the use of a microneedle (Sunlight Medical, Jacksonville, FL, USA) and transferred in a 10 % polyvinylpyrrolidone (PVP) solution (SAGE, USA), immobilized, and then used to inject sibling MII oocytes. The procedure was carried out under an inverted microscope equipped with a holding pipette with slight negative pressure for handling the oocyte and an injection needle for injecting the sperm. The immature oocytes used for sperm selection were discarded. In all groups, the injection needle containing a single sperm was steadily and slowly moved through the cytoplasm of the MII oocyte and dropped 1 to 3µl to the center of the oocyte .

6- Outcome measures: All the embryological parameters (i.e. fertilization, cleavage, blastocyst formation, and blastocyst quality) were recorded and assessed. Signs for fertilization were observed 16-18 hours post ICSI. Furthermore, 48 and 72 h after ICSI, the cleavage rate was assessed. The blastocyst formation rate was assessed on day five post-ICSI. Embryos with high-quality blastocyst formation were classified according to Gardner's blastocyst grading system. This system assigns grades of the expansion and hatching status according to inner cell mass (ICM) and the trophectoderm (TE) quality. Good-quality blastocysts were classified as those with 6, 5, 4, or 3AA, AB, or BA. Fair-quality blastocysts were those with 6, 5, 4, or 3 BB.

7-Statistical analysis The rates of fertilization, cleavage, blastocyst formation, and high-quality blastocysts were reported as percentages for each group. Characteristics of male and female patients (age, sperm count, sperm motility, sperm morphology, number of retrieved oocytes, and number of mature and immature oocytes) were expressed as mean ± standard deviation (SD). The Student t-test was employed to compare continuous variables (fertilization rates, cleavage, blastocyst formation, and high-quality blastocysts). Statistical analysis was performed with SPSS 13.0. P-value ≤ 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Couples must be diagnosed with infertility and undergoing ICSI cycle.
* The age range for all female subjects must be between 21 and 38 years old, and their male partners must be older than 24 years old and above 50 years old.
* Patients must produce at least two mature oocytes (one to be used for control and one for treatment) and one immature oocyte (to be used for selecting sperm).
* Males must show at least 10% total sperm motility

Exclusion Criteria:

* Cases where the female was younger than 21 years or older than 38 years old.
* Patients that had less than two mature oocytes
* Patients with no immature oocytes
* Patients with low oocyte quality.
* Cases with less than 10% motility or those with no motility such as PESA, TESA, and TESE cases.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
fertilization rate | 17-18 hours post ICSI
  percentage of transformation of micro injected oocytes into two pronuclei
cleavage rate | 44 ± 1 h post ICSI
  percentage of cleavage of fertilized oocytes into 2-4 cell embryos
high-quality cleaved embryos rate | 68 ± 1 h post ICSI
  percentage of total number of high-quality day-3 embryos by total number of cleaved embryos
blastocyst formation rate | 107.9-112.9 hours after ICSI
  percentage of total number of embryos transformed into blastocysts by total number of cleaved embryos
high-quality blastocyst rate | 107.9-112.9 hours after ICSI
  percentage of total number of high-quality expanded blastocysts on day 5 and/or 6 by total number of blastocysts

CONTACTS AND LOCATIONS:
Overall Officials: Nehal A Abu Elnaga, PhD, Study Director — Al-Azhar University
Locations (1):
- Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No